CLINICAL TRIAL: NCT03353142
Title: The Effects Of Equal Breathing On Pain Pressure Thresholds In Individuals With Chronic Low Back Pain: A Pilot Study
Brief Title: The Effects Of Equal Breathing On Pain Pressure Thresholds
Acronym: EB-Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hamilton Health Sciences Corporation (Other)
Responsible Party: Principal Investigator, Gurpreet Palak, Physician - Fellow, Hamilton Health Sciences Corporation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MGD-004-20171016
Record Dates: First submitted 2017-11-06; First posted 2017-11-27 (Actual); Last update posted 2018-06-14 (Actual); Status verified 2018-06

CONDITIONS: Chronic Low Back Pain

STUDY DESIGN:
Intervention Model Description: Consecutive participants meeting eligibility criteria will be enrolled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Equal Breathing (Experimental)
  Interventions: Other: Equal Breathing

INTERVENTIONS:
Other: Equal Breathing — * Blood pressure recorded at baseline, immediately pre- and post-trial
  * Maximum Tolerable Breathing Ratio: Test run to determine the maximum tolerable time for inhalation and exhalation.
  * PRESSURE TOLERANCE: Pressure algometer device used to determine pain pressure tolerance. It will be applied to the first dorsal interosseous and deltoid, and pain pressure tolerance will be measured and recorded. Pressure will be applied at 1kg per second until the patient indicates that the pressure has become painful. Pain pressure tolerance will be performed 3 times at each anatomical location and an average will be determined for each location.
  * TRIAL: Participants will begin 5 minutes of Equal Breathing at their maximum tolerable equal breathing ratio that was previously determined. Immediately after 5 minutes of breathing, the pain pressure tolerance will be measured using pressure algometry

SUMMARY:
Recent research has found that there is moderate evidence for the use of breathing exercises for treating chronic, non-specific low back pain. Researchers have found that there were significant improvements in pain and quality of life in those suffering with low back pain who completed a breathing program intervention. Researchers also found that healthy individuals had higher pain thresholds and tolerance following deep and slow breathing exercises.

There are numerous formats of breathing interventions, some interventions that have been used with individuals with chronic, non-specific low back pain include: deep breathing, yoga breathing, resisted inspiration, and breathe holding. There is moderate evidence to suggest the use of these interventions for managing chronic low back pain Another common breathing format is Equal-Ratio Breathing. This format requires an individual to inhale and exhale with the same duration while gradually increasing the duration of both. This breathing format can be easier for patients to perform given the simplicity of the equal inhalation to exhalation ratio.

This research is being done because Equal-Ratio Breathing has yet to be studied in individuals with chronic low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18
* Chronic low back pain
* OHIP patient

Exclusion Criteria:

* Peripheral pain
* Peripheral neuropathy
* Chronic regional pain syndrome
* Alpha and Beta blocker medication use
* Patient does not wish to participate
* Completed or participated in a psychoeducational program at the clinic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-02-01 (Estimated); Study Completion 2019-02-01 (Estimated)

PRIMARY OUTCOMES:
Difference in pain pressure threshold | Pre-visit and Post-visit - same day
  Measured using the pressure algometer device

SECONDARY OUTCOMES:
Difference in heart rate | Pre-visit and Post-visit - same day
  Measure by pulse oximeter
Difference in blood pressure values | Pre-visit and Post-visit - same day
  Measure by pulse oximeter

CONTACTS AND LOCATIONS:
Locations (1):
- Michael G. DeGroote Pain Clinic, Hamilton Health Sciences, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
no plan to share IPD